CLINICAL TRIAL: NCT00792415
Title: Validation of a Pediatric Abstinence Syndrome Scoring Tool Utilizing a Standardized Hospital-Based Guideline for Iatrogenic Opioid Dependence
Brief Title: Validation of a Pediatric-Specific Abstinence Syndrome Assessment Tool
Status: Withdrawn | Type: Observational
Why Stopped: Study doctor no longer with Banner Health, please remove this study from our list.
Sponsor: Banner Health (Other)
Responsible Party: Sponsor
Other Study IDs: BHRI#05-08-0074
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Substance Withdrawal Syndrome
Keywords: Abstinence syndrome symptoms; Withdrawal symptoms; Opioid dependence
MeSH Terms: conditions — Substance Withdrawal Syndrome; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the validity and reliability of an abstinence syndrome assessment tool used in pediatric patients with iatrogenic opioid dependence.

DETAILED DESCRIPTION:
None available.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Intensive Care Unit patients ages 2 weeks to 18 years
* Patients receiving continuous opioid infusions for 5 days (at least 120 hours) or more

Exclusion Criteria:

* Attending discretion
* Patients with deterioration of medical status requiring interventions of pain control, surgery, sedation, or re-intubation

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Intensive Care Unit patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Total scores of abstinence syndrome symptoms | Up to 23 days
  None available - PI no longer with Banner

SECONDARY OUTCOMES:
Expert opinion on abstinence syndrome | Up to 23 days
  None available - PI no longer with Banner

CONTACTS AND LOCATIONS:
Overall Officials: Teri Reyburn-Orne, RN, MSN, PNP, Principal Investigator — Banner Children's Hospital at Banner Desert Medical Center
Locations (1):
- Cardon Children's Medical Center, Mesa, Arizona, United States